CLINICAL TRIAL: NCT05176951
Title: A Phase 2, Randomized, Double-Blind, Multicenter, Placebo-Controlled Study to Evaluate the Safety and Tolerability of Treprostinil Palmitil Inhalation Powder in Participants With Pulmonary Hypertension Associated With Interstitial Lung Disease
Brief Title: A Study to Evaluate the Safety and Tolerability of Treprostinil Palmitil Inhalation Powder in Participants With Pulmonary Hypertension Associated With Interstitial Lung Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INS1009-211; 2021-003294-66 (EudraCT Number)
Record Dates: First submitted 2021-12-10; First posted 2022-01-04 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Interstitial Lung Disease; Treprostinil Palmitil
MeSH Terms: conditions — Hypertension, Pulmonary; Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treprostinil Palmitil (Experimental): Participants will be administered TPIP once per day at a starting dose of 80 micrograms (μg). Participants will be titrated up to the highest tolerated dose for each individual participant of between 80 μg and 640 μg during the initial 3 weeks of treatment. The overall treatment period will be 16 weeks.
  Interventions: Drug: Treprostinil Palmitil
- Placebo (Placebo Comparator): Participants will be administered a placebo matching TPIP once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Treprostinil Palmitil — Oral inhalation using a capsule-based dry powder inhaler device.
  Other Names: INS1009
  Arms: Treprostinil Palmitil
Drug: Placebo — Oral inhalation using a capsule-based dry powder inhaler device.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of treprostinil palmitil inhalation powder (TPIP) compared with placebo

ELIGIBILITY:
Inclusion Criteria:

* Males and females must be ≥ 18 to ≤ 80 years of age at the time of signing the informed consent form (ICF).
* Diagnosis of pulmonary hypertension (PH) associated with interstitial lung disease (ILD) (including idiopathic interstitial pneumonia [IIP], idiopathic pulmonary fibrosis [IPF], connective tissue disease [CTD], sarcoidosis).
* Male and female participants must use contraceptives that are consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Male participants:

Male participants who are not sterile, with female partners of childbearing potential, must be using effective contraception from Day 1 to at least 90 days after the last dose of study drug.

Male participants with women of child bearing potential (WOCBP) partner must use a condom in order to avoid potential exposure to embryo/fetus.

- Female participants: Women must be postmenopausal (defined as no menses for 12 months without an alternative medical cause), surgically sterile, (ie,hysterectomy and/or bilateral salpingo-oophorectomy) or using highly effective contraception methods (ie, methods that alone or in combination achieve <1% unintended pregnancy rates per year when used consistently and correctly) from Day 1 to at least 90 days after the last dose of study drug.

- Capable of giving signed informed consent that includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

* Primary diagnosis of chronic obstructive pulmonary disease (COPD).
* Allergy, or documented hypersensitivity or contraindication to TPIP or treprostinil (TRE) or mannitol (an excipient of the TPIP formulation).
* Received or currently treated with riociguat, endothelin receptor antagonists, selexipag, phosphodiesterase 5 (PDE5) inhibitors and/or prostacyclin analogues within 30 days prior to Screening.
* Started therapy with pirfenidone or nintedanib < 90 days prior to Screening, OR, if already receiving either medication, there is a dose change within 30 days of Screening Visit.
* Any known ventricular or supraventricular tachyarrhythmia (except for paroxysmal atrial fibrillation), and/or any symptomatic bradycardia.
* History of heart disease including left ventricular ejection fraction (LVEF) ≤ 40% or clinically significant valvular, constrictive, or symptomatic atherosclerotic heart disease (eg, stable angina, myocardial infarction, etc).
* Participation in a cardiopulmonary rehabilitation program within 30 days of the first Screening Visit. Participation in the maintenance program of a cardiopulmonary rehabilitation program is allowed.
* Acutely decompensated heart failure within 30 days of Screening Visit.
* Active and current symptomatic coronavirus disease 2019 (COVID-19) and/or previous diagnosis of moderate to severe disease, or hospitalization due to COVID-19.
* Supplemental oxygen requirement > 10L/min at rest at Screening.
* Exacerbation of underlying lung disease or active pulmonary or upper respiratory infection within 30 days of the first dose of study drug (may be rescreened at appropriate time).
* Current or recent (past 30 days) lower respiratory tract infection (may be rescreened at appropriate time).
* Any form of congenital heart disease or congenital heart defect (repaired or unrepaired) other than a patent foramen ovale.
* History of alcohol or drug abuse within 6 months prior to Screening.
* Current use of cigarettes (as defined by Center for Disease Control (CDC)) or e-cigarettes: An adult who has smoked at least 100 cigarettes in his or her lifetime and who currently smokes either every day or some days.
* Participants who currently inhale marijuana (recreational or medical).
* Acute or chronic impairment (other than dyspnea), limiting the ability to comply with study requirements, in particular with 6-minute walk test (6MWT) (eg, angina pectoris, claudication, musculoskeletal disorder, need for walking aids).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experience Any Number of Treatment Emergent Adverse Events (TEAEs) | Up to Day 140
Number of Participants Who Experience Any Number of Serious Adverse Events (SAEs) | Up to Day 140
Change from Baseline in Saturation of Peripheral Capillary Oxygenation (SpO2) Levels | Pre-, during, and post- 6-minute walk test (6MWT) at Baseline, Week 5, Week 10, and Week 16

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Treprostinil Palmitil | Day 1 to Week 16
Cmax of Treprostinil | Day 1 to Week 16
Time to Maximum Plasma Concentration (Tmax) of Treprostinil Palmitil | Day 1 to Week 16
Tmax of Treprostinil | Day 1 to Week 16
Area Under Concentration-time Curve From Time 0 to 24 Hours Post-dose (AUCtau) of Treprostinil Palmitil | Day 1 to Week 16
AUCtau of Treprostinil | Day 1 to Week 16
Area Under Concentration-time Curve From 0 to Infinity (AUC∞) of Treprostinil Palmitil | Day 1 to Week 16
AUC∞ of Treprostinil | Day 1 to Week 16
Area Under Concentration-time Curve From Time 0 to Last Measurable Concentration (AUClast) of Treprostinil Palmitil | Day 1 to Week 16
AUClast of Treprostinil | Day 1 to Week 16
Apparent Total Clearance (CL/F) of Treprostinil Palmitil | Day 1 to Week 16
CL/F of Treprostinil | Day 1 to Week 16
Elimination Half-life (t1/2) of Treprostinil Palmitil | Day 1 to Week 16
t1/2 of Treprostinil | Day 1 to Week 16
Apparent Volume of Distribution After Terminal Phase (Vd/F) of Treprostinil Palmitil | Day 1 to Week 16
Vd/F of Treprostinil | Day 1 to Week 16

CONTACTS AND LOCATIONS:
Locations (25):
- Argentina (3):
  - ARG003, Barracas, Ciudad Autónoma de BuenosAires
  - ARG001, Rosario, Santa Fe Province
  - ARG008, Buenos Aires
- Australia (2):
  - AUS003, Camperdown, New South Wales
  - AUS005, Macquarie Park, New South Wales
- BEL002, Liège, Belgium
- Germany (7):
  - GER006, Heidelberg, Baden-Wurttemberg
  - GER010, Giessen, Hesse
  - GER003, Essen, North Rhine-Westphalia
  - GER001, Dresden, Saxony
  - GER002, Berlin
  - GER012, Berlin
  - GER004, Munich
- Italy (4):
  - ITA003, Napoli, Campania
  - ITA004, Milan, Lombardy
  - ITA002, Monza, Lombardy
  - ITA001, Palermo, Sicily
- Spain (6):
  - ESP003, Palma de Mallorca, Balearic Islands
  - ESP007, Oviedo, Principality of Asturias
  - ESP010, Barcelona
  - ESP005, Barcelona
  - ESP006, Las Palmas de Gran Canaria
  - ESP009, Santiago de Compostela
- United Kingdom (2):
  - GBR003, Glasgow, Lanarkshire
  - GBR001, Sheffield, Yorkshire

IPD SHARING:
Plan to Share IPD: No